CLINICAL TRIAL: NCT01861210
Title: Couples HIV Counseling and Testing for Male Couples in the United States
Acronym: CVCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Patrick S Sullivan, Professor, Emory University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00043714; R34MH086331 (NIH); CVCTMSM (Other: Other)
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: HIV
Keywords: Homosexuality, Male
MeSH Terms: conditions — Homosexuality, Male | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Couples Counseling and Testing (Experimental): Couples Voluntary HIV Counseling and Testing, adapted for use with male couples from the standard African couples testing service.
  Interventions: Behavioral: Couples Voluntary HIV Counseling and Testing
- Individudal Counseling and Testing (Active Comparator): Individual Voluntary Counseling and Testing involves HIV testing and individual, client-centered HIV prevention counseling. This service is provided by counselors trained in Centers for Disease Control and Prevention's "Fundamentals of HIV Prevention Counseling" training.
  Interventions: Behavioral: Individual Counseling and Testing

INTERVENTIONS:
Behavioral: Couples Voluntary HIV Counseling and Testing
  Other Names: Couples HIV Testing and Counseling
  Arms: Couples Counseling and Testing
Behavioral: Individual Counseling and Testing
  Arms: Individudal Counseling and Testing

SUMMARY:
This is a study to determine whether testing for HIV together as a couple, as opposed to testing separately, in acceptable to men in male couples, and is a safe prevention service. Testing of couples together has been provided for decades in Africa, but has never been tested in the United States. In this study, male couples will be enrolled and randomly assigned to be tested together in the same room, or separately. At the time of testing, investigators will ask questions about how they felt about the service they received. Three months later, investigators will survey the men again, and determine whether they had any problems after the testing, like violence in the relationship or the relationship breaking up. The main outcomes are being satisfied with the testing service, and safety (lack of intimate partner violence or relationship termination). Although the study is not designed to determine if the service reduces risk behaviors for HIV transmission, investigators will examine data on risks just to explore that topic. The main hypotheses are: (1) men will be at least as satisfied with couples testing as they are with individual testing; and (2) men tested as couples will not experience higher rates of intimate partner violence or relationship dissolution, relative to men tested separately.

ELIGIBILITY:
Inclusion Criteria:

* male at birth
* currently self-identify as male
* at least 18 years of age
* have been in a couple with a man for at least 3 months
* willing to complete a follow-up study visit in 3 months
* able to complete study assessments in English.

Exclusion Criteria:

* known to be HIV-positive
* over 39 years of age
* either partner being unwilling to accept randomization to the couples testing arm
* either partner planning to move from the Atlanta area within 3 months of the initial study visit
* either partner reporting a history of intimate partner violence
* either partner reporting feeling coerced to tested with his partner

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2010-09; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Intimate partner violence | 3 months
  Having been punched, hit, or kicked by the partner he tested with, injured to the point of feeling physical pain the day after a fight, or inflicting any of these acts on his partner in the preceding three months.

SECONDARY OUTCOMES:
Relationship dissolution | 3 months, or at the time of followup survey
  Either or both partners reported that the relationship ended after their participation in the study

OTHER OUTCOMES:
Satisfaction with counseling service | Within 30 minutes after the service
  Seven items asked on a 5-point Likert scale:
  * Quality of the session
  * Relevance of the session
  * Appropriateness of the format
  * Degree to which the session met personal needs
  * Usefulness of the session
  * Satisfaction with the session
  * Likelihood of recommending the service to a friend

CONTACTS AND LOCATIONS:
Overall Officials: Patrick S Sullivan, PhD, Principal Investigator — Emory University Rollins School of Public Health
Locations (1):
- AID Atlanta, Atlanta, Georgia, United States